CLINICAL TRIAL: NCT01780519
Title: The Cognitive Effects of Lorazepam in Healthy Older Individuals With TOMM40 Variable-length Polymorphisms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Cynthia M. Stonnington, M.D., PI, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 12-006469
Record Dates: First submitted 2013-01-29; First posted 2013-01-31 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Alzheimer's Disease (AD)
Keywords: Alzheimer's disease (AD)
MeSH Terms: conditions — Alzheimer Disease | interventions — Lorazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- L/VL APOE e3/e4 carrier (Other): long and very long poly - T variants of TOMM40 and APOE e3/e4 carrier
  Interventions: Drug: lorazepam
- L/S APOE e3/e4 carrier (Other): long and short poly - T variants of TOMM40 and APOE e3/e4 carrier
  Interventions: Drug: lorazepam
- S/VL APOE e3/e3 carrier (Other): short and Very long poly - T variants of TOMM40 and APOE e3/e3 carrier
  Interventions: Drug: lorazepam
- VL/VL APOE e3/e3 carrier (Other): Very long poly - T variants of TOMM40 and APOE e3/e3 carrier
  Interventions: Drug: lorazepam
- S/S APOE e3/e3 carrier (Other): short poly - T variants of TOMM40 and APOE e3/e3 carrier
  Interventions: Drug: lorazepam

INTERVENTIONS:
Drug: lorazepam — single dose of 1 mg lorazepam
  Other Names: Ativan

SUMMARY:
The investigators' goal is to determine if certain tests of memory and attention, performed while sleepiness is induced by a single dose of lorazepam, can predict whether or not an individual is at risk for developing Alzheimer's disease.

ELIGIBILITY:
Inclusion criteria:

* Mini-Mental State Examination (MMSE) score of 28-30
* Hamilton Depression Rating Scale score of less than 10
* participants in longitudinal study of aging and have a TOMM40 genotype of S/S, VL/VL, S/VL, L/S or L/VL.

Exclusion criteria:

* Alzheimer's Disease or Mild Cognitive Impairment
* any significant medical, psychiatric, and neurological illnesses, e.g., impaired liver or kidney function, prior stroke, traumatic brain injury, memory impairment, cognitive impairment, parkinsonism, a lifetime history of schizophrenia, bipolar disorder, a psychoactive substance use disorder, or current major depression.
* known allergy to benzodiazepines
* current use (within the previous four weeks) of benzodiazepines or other medications known to interact with lorazepam, current use of sedating antihistamines, or current use of stimulant medications

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Groton Maze Learning Test (GMLT) score | baseline to 5 hours
  The GMLT assesses visuospatial working memory, error monitoring, information processing speed, and short-term delayed recall for a complex hidden maze. Subjects are familiarized with the task during two untimed practice tests, and once the tester is confident that the subject understands the rules and can move easily around the grid, the timed test is administered. In each of the 5 successive trials of the GMLT exam, the subject is asked to learn to navigate his or her way around a 28-step maze that is hidden beneath a 10 x 10 grid of squares on the computer touch screen. For each trial, the time to completion, number of correct moves, number of wrong moves, and the number of perseverative errors are recorded.

SECONDARY OUTCOMES:
Auditory Verbal Learning Test (AVLT) Long-term memory score | baseline to 5 hours
  The AVLT assesses verbal memory
Two Back Test (TBK) | baseline to 5 hours
  The TBK measures working memory

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Stonnington, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Scottsdale, Arizona, United States